CLINICAL TRIAL: NCT03595709
Title: Prospective, Therapeutic Drug Monitoring Study of Reduced-Dose Efavirenz (400 mg) Plus Tenofovir Disoproxil Fumarate (TDF) and Lamivudine in a Fixed-Dose Combination Tablet (Combo) for Patients Receiving Co-Formulated TDF, Emtricitabine and Efavirenz (Atripla) With Viral Suppression in Taiwan
Brief Title: Therapeutic Drug Monitoring Study of Reduced-Dose Efavirenz (400 mg) in Combo Tablet for Patients Receiving Atripla With Viral Suppression in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yu-Jay Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YJ14001-COMBO-201801
Record Dates: First submitted 2018-07-02; First posted 2018-07-23 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections
Keywords: Efavirenz; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined tablet (EFV 400,TDF 300, 3TC 300) (Experimental): All eligible subjects will receive 3-in-1 tablet (EFV 400mg, TDF 300mg, 3TC 300mg) once daily for 24 weeks orally on empty stomach before bedtime. If the event of toxicity or tolerability issues requires a change from study drug, switching to the best available treatment will be recommended.
  Interventions: Drug: 3-in-1 tablet (EFV 400mg, TDF 300mg, 3TC 300mg)

INTERVENTIONS:
Drug: 3-in-1 tablet (EFV 400mg, TDF 300mg, 3TC 300mg) — All eligible subjects will receive 3-in-1 tablet (EFV 400mg, TDF 300mg, 3TC 300mg) once daily for 24 weeks orally on empty stomach before bedtime. If the event of toxicity or tolerability issues requires a change from study drug, switching to the best available treatment will be recommended.
  Other Names: non applicable

SUMMARY:
Prospective, Therapeutic Drug Monitoring Study of Reduced-Dose Efavirenz (400 mg) Plus Tenofovir Disoproxil Fumarate (TDF) and Lamivudine in a Fixed-Dose Combination Tablet (Combo) for Patients Receiving Co-Formulated TDF, Emtricitabine and Efavirenz (Atripla) with Viral Suppression in Taiwan

DETAILED DESCRIPTION:
Efavirenz (EFV) is the most widely used non-nucleoside reverse transcriptase inhibitor (NNRTI). The recommended dose of EFV is 600 mg daily; however, a phase II study showed no significant difference in viral suppression rates across the different EFV groups (200 mg, 400 mg, and 600 mg) at 24 weeks. The week 96 analysis of ENCORE 1 study confirmed the durable virological non-inferiority of EFV 400 mg to the standard 600 mg dose when given as initial therapy with tenofovir disoproxil fumarate (TDF) and emtricitabine (FTC). Fewer EFV-related adverse events (AEs) and fewer treatment discontinuations were also observed in the reduced dose group. The efficacy and safety findings provide robust evidence to redefine the EFV dose for HIV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving co-formulated TDF/ FTC/ EFV (600 mg) and have achieved an undetectable plasma viral load (<50 copies/mL) for 6 months or longer at screening visit.
* Having C12 EFV of 1 mg/L or greater at screening.
* (C12 EFV will be determined by using blood sample collected 12 ± 1 hour after previous dosing of co-formulated TDF/ FTC/ EFV (600 mg).
* No known treatment failure to regimens containing TDF, 3TC or FTC, plus EFV.
* Infected with HIV harboring no known resistance-associated mutations to EFV, TDF, 3TC or FTC.
* No known allergies to EFV, TDF, 3TC or FTC.
* Aged ≧20 years.
* Calculated creatinine clearance (ClCr) ≥ 50 mL/min (Cockcroft-Gault formula).
* Provision of written informed consent.

Exclusion Criteria:

* The following laboratory values:

  * Absolute neutrophil count (ANC) <500 cells/μL
  * Hemoglobin <7.0 g/dL
  * Platelet count <50,000 cells/μL
  * Serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >5x upper limit of normal (ULN)
* Pregnant women or nursing mothers.
* Active opportunistic or malignant disease not under adequate control.
* Use of immunomodulators within 30 days prior to screening visit.
* Use any of the prohibited medications: bepridil, astemizole, terfenadine, dihydroergotamine, ergometrine, ergotamine, systemic cytotoxic chemotherapy, amodiaquine, pimozide, midazolam, triazolam, cisapride、St John's Wort、 Elbasvir/Grazoprevir and Simeprevir.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
C12 EFV concentration | Week 4
  The proportion of subjects achieving C12 EFV concentration >1.0 mg/L at Week 4.

SECONDARY OUTCOMES:
HIV-1 RNA load | Week 12
  The proportion of subjects with undetectable plasma HIV-1 RNA load (<50 copies/mL) at Week 12
HIV-1 RNA load | Week 24
  The proportion of subjects with undetectable plasma HIV-1 RNA load (<50 copies/mL) at Week 24
EFV concentration | Week 4
  The mean changes from baseline in C12 EFV concentration at Week 4.
CD4+ T cell count | Week 12
  The mean changes from baseline in CD4+ T cell count at Week 12.
CD4+ T cell count | Week 24
  The mean changes from baseline in CD4+ T cell count at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yun Sun, MD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - E-Da Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No